CLINICAL TRIAL: NCT03322865
Title: Obinutuzumab in Marginal Zone Lymphoma (OLYMP-1)
Brief Title: Obinutuzumab in Marginal Zone Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Christian Buske (Other)
Collaborators: University of Ulm (Other); Optimapharm (Industry); Zentrum für Klinische Studien Ulm (Other); X-act Cologne Clinical Research GmbH (Industry); Roche Pharma AG (Industry)
Responsible Party: Sponsor-Investigator, Christian Buske, Prof. Dr. med., University of Ulm
Organization: University of Ulm (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OLYMP-1; 2017-003149-56 (EudraCT Number)
Record Dates: First submitted 2017-10-11; First posted 2017-10-26 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Marginal Zone Lymphoma
Keywords: Obinutuzumab; Anti-CD20 antibody; Oncology
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Neoplasms | interventions — obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- One Arm (Experimental): Obinutuzumab i.v.
  Interventions: Drug: Obinutuzumab

INTERVENTIONS:
Drug: Obinutuzumab — Induction:
  Cycle 1 (28 days cycle): Obinutuzumab (OBINUTUZUMAB) 1000mg i.v. fixed dose day 1,8,15*
  *In the case of suspected increased risk of severe IRR, the dose of obinutuzumab may be 100 mg intravenously on day 1 in cycle 1, 900 mg on day 2.
  Cycle 2-6 (28 days cycle): Obinutuzumab (OBINUTUZUMAB) 1000mg i.v. fixed dose day 1 Maintenance
  Start 8 weeks after the last induction cycle for patients at least achieving a partial response after induction:
  Obinutuzumab (OBINUTUZUMAB) 1000mg i.v. fixed dose day 1 every 8 weeks for a maximum of 12 infusions unless progression or study drug - related intolerable toxicity
  Other Names: GA101

SUMMARY:
For marginal zone lymphoma (MZL) Rituximab in combination with conventional chemotherapy are widely used for those patients who fail local therapy or do not qualify for such. Depending on the MZL subtype Rituximab/chemotherapy is able to induce in part long remissions, but do not prevent relapse later on. In addition, chemotherapy associated toxicity is often problematic in MZL patients, who are mostly of advanced age. Thus, chemotherapy - free approaches are highly attractive for this patient group. Rituximab single agent is a widely used chemotherapy - free approach in MZL, but was significantly inferior compared to Rituximab/chlorambucil in a large randomized prospective clinical trial in treatment naïve MZL with a CR rate of 56 % vs. 80%, respectively (P<0.001).Thus, it is the major aim to develop chemotherapy - free approaches for MZL, which approach efficacy of rituximab/chemotherapy combinations, but avoid chemotherapy associated toxicities. This in particular important in MZL as many physicians are reluctant to treat these often elderly patients with more intense treatments and prefer single agent therapies in these very often well and long responding lymphoma subtype. The type II anti-CD20 antibody Obinutuzumab (OBINUTUZUMAB) has demonstrated remarkable activity in follicular lymphoma and superiority to Rituximab in combination with chemotherapy in treatment naïve (Gallium trial) and rituximab refractory follicular lymphoma (Gadolin trial) as well as in CLL in combination with chlorambucil. Based on these observations it is the aim of this study to test the toxicity and efficacy of the anti-CD20 antibody Obinutuzumab (OBINUTUZUMAB) in patients with newly diagnosed MZL in need of treatment, who are not eligible or failed local therapy, following the assumption that this novel anti-CD20 antibody is significantly more effective than Rituximab single agent therapy, and avoids chemotherapy - related toxicity.

DETAILED DESCRIPTION:
For marginal zone lymphoma (MZL) Rituximab in combination with conventional chemotherapy are widely used for those patients who fail local therapy or do not qualify for such. Depending on the MZL subtype Rituximab/chemotherapy is able to induce in part long remissions, but do not prevent relapse later on. In addition, chemotherapy associated toxicity is often problematic in MZL patients, who are mostly of advanced age. Thus, chemotherapy - free approaches are highly attractive for this patient group. Rituximab single agent is a widely used chemotherapy - free approach in MZL, but was significantly inferior compared to Rituximab/chlorambucil in a large randomized prospective clinical trial in treatment naïve MZL with a CR rate of 56 % vs. 80%, respectively (P<0.001).Thus, it is the major aim to develop chemotherapy - free approaches for MZL, which approach efficacy of rituximab/chemotherapy combinations, but avoid chemotherapy associated toxicities. This in particular important in MZL as many physicians are reluctant to treat these often elderly patients with more intense treatments and prefer single agent therapies in these very often well and long responding lymphoma subtype. The type II anti-CD20 antibody Obinutuzumab (OBINUTUZUMAB) has demonstrated remarkable activity in follicular lymphoma and superiority to Rituximab in combination with chemotherapy in treatment naïve (Gallium trial) and rituximab refractory follicular lymphoma (Gadolin trial) as well as in CLL in combination with chlorambucil. Based on these observations it is the aim of this study to test the toxicity and efficacy of the anti-CD20 antibody Obinutuzumab (OBINUTUZUMAB) in patients with newly diagnosed MZL in need of treatment, who are not eligible or failed local therapy, following the assumption that this novel anti-CD20 antibody is significantly more effective than Rituximab single agent therapy, and avoids chemotherapy - related toxicity. For efficacy the rate of complete remissions (according to the GELA criteria for gastric MALT or to the Cheson 2007 criteria for non-gastric extranodal, nodal and splenic MZL) after induction therapy will be primarily analysed. For toxicity treatment associated adverse events, quality of life and cumulative incidence of secondary malignancies will be documented.

The study is a multicenter, single-arm, open-label, phase II trial of 6 cycles of Obinutuzumab in the induction phase followed by a maintenance phase for a maximum of 12 infusions of Obinutuzumab every 8 weeks in patients aged ≥ 18 years with previously untreated MZL in need of treatment.

The study flow will be as follows:

* Previously untreated patients will be screened for eligibility for the trial. If the patient is eligible for the study, the patient will be registered before the first cycle of induction treatment.
* Patients who progress at any time point during induction are considered as treatment failure. They will be followed up for overall survival until death.
* Patients, who achieve at least a SD after induction treatment will be eligible to receive maintenance therapy with Obinutuzumab.

It is expected that a total of 56 patients at approximately 20 investigator sites will be registered. Every patient will receive treatment over a time period of 6 x 4 weeks, followed by a maintenance phase of every 8 weeks for a maximum of 12 infusions until progression or study drug - related intolerable toxicity. Patient will be monitored every 3 months for 2 additional years, subsequently every 6 months for three additional years.

ELIGIBILITY:
Inclusion Criteria:

Patients must have a proven pathological diagnosis of MZL.

Patients must meet all of the following inclusion criteria to be eligible for participation in this study:

* Confirmed CD20 positive de novo MALT Lymphoma following or being not eligible for local therapy (including surgery, radiotherapy) and antibiotics for H. pylori-positive gastric lymphoma arisen at any extranodal site
* Confirmed CD20 positive de novo splenic MZL following or not being eligible for local therapy (including surgery and antiviral therapy for Hepatitis C Virus) with symptomatic disease
* Confirmed CD20 positive de novo nodal MZL
* Patients in need of treatment:

For patients with symptomatic splenic, nodal, or non-gastric extranodal MZL disease that is de novo or has relapsed following local therapy (i.e., surgery or radiotherapy) and requires therapy, as assessed by the investigator.

For patients with symptomatic gastric extranodal MZL: Helicobacter pylori-negative disease that is de novo or has relapsed following local therapy (i.e., surgery or radiotherapy) and requires therapy, as assessed by the investigator, or H. pylori-positive disease that has remained stable, progressed, or relapsed following antibiotic therapy and requires therapy, as assessed by the investigator - At least one bi-dimensionally measurable lesion (> 2 cm in its largest dimension by CT scan or MRI).

In patients with splenic MZL, an enlarged spleen on CT scan or extending at least 2 cm below the costal margin by physical examination will constitute measurable disease providing that no explanation other than lymphomatous involvement is likely. For an enlarged liver to constitute the only measurable disease parameter, a liver biopsy showing proof of NHL in the liver is required.

For SMZL:

* Bulky progressive or painful splenomegaly
* one of the following symptomatic/progressive cytopenias : Hb < 10 g/dL, or Plat < 80.000 /microL, or neutropenia < 1000 /microL, whatever the reason (autoimmune or hypersplenism or bone marrow infiltration)
* enlarged lymphoadenopathy or involvement of extranodal sites with or without cytopenia
* splenectomised patients with rapidly raising lymphocyte counts, development of lymphadenopathy or involvement of extranodal sites
* SMZL with concomitant hepatitis C infection who have not responded to or are relapsed after Interferon and/or Ribavirin (patients positive for HCV antibody are eligible only if PCR is negative for HCV RNA.

For gastric MALT Lymphoma:

- H. pylori-negative cases following or being not eligible for local therapy (i.e., surgery, radiotherapy or antibiotics).

Others:

* Age greater than 18 years
* Life expectancy >3 months.
* Baseline platelet Count 50, 109/L, if not due to BM Infiltration by the lymphoma, absolute neutrophil Count 0.75, 109/L
* Meet the following pretreatment laboratory criteria at the Screening visit conducted within 28 days of study enrollment (unless due to underlying lymphoma):
* ASAT (SGOT): 3 times the upper limit of institutional laboratory normal value
* ALAT (SGPT): 3 times the upper limit of institutional laboratory normal value
* Total Bilirubin: 20 mg/L or 2 times the upper limit of institutional laboratory normal value, unless clearly related to the disease (except if due to Gilbert's syndrome)
* Serum creatininie <= 2mg/dl
* Pregnancy beta-HCG negative. For women of child-bearing potential only; serum or urine beta-HCG must be negative during screening and at study enrolment visit
* Negative HIV antibody
* Positive test results for chronic HBV infection (defined as positive HBsAg serology): patients with occult or prior HBV infection (defined as negative HBsAg and positive total HBcAb) may be included if HBV DNA is undetectable, provided that they are willing to undergo monthly DNA testing. Patients who have protective titers of HBSAb after vaccination or prior but cured hepatitis B are eligible.
* Positive test results for hepatitis C (hepatitis C virus (HCV) antibody serology testing): patients positive for HCV antibody are eligible only if PCR is negative for HCV RNA.
* Premenopausal fertile females must agree to use a highly effective method of birth control for the duration of the therapy up to 6 months after end of therapy. A highly effective method of birth control is defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some IUDs, sexual abstinence or vasectomised partner.
* Men must agree not to father a child for the duration of therapy and 6 months after and must agree to advice a female partner to use a highly effective method of birth control.
* Willingness and ability to comply with scheduled visits, drug administration plan, imaging studies, laboratory tests, other study procedures, and study restrictions.
* Evidence of a personally signed informed consent indicating that the subject is aware of the neoplastic nature of the disease and has been informed of the procedures to be followed, the experimental nature of the therapy, alternatives, potential benefits, possible side effects, potential risks and discomforts, and other pertinent aspects of study participation.

The presence of any of the following will exclude a subject from enrolment:

* ECOG performance status >2
* History of a non-lymphoid malignancy except for the following: adequately treated local basal cell or squamous cell carcinoma of the skin, cervical carcinoma in situ, superficial bladder cancer, asymptomatic prostate cancer without known metastatic disease and with no requirement for therapy or requiring only hormonal therapy and with normal prostate specific antigen for ≥1 year prior to study enrollment visit, other Stage 1 or 2 cancer treated with a curative intent and currently in complete remission, for ≥3 years.
* Central nervous system lymphoma, leptomeningeal lymphoma, or histologic evidence of transformation to a high-grade or diffuse large B-cell lymphoma.
* Ann Arbor Stage I disease
* Ongoing immunosuppressive therapy other than corticosteroids
* Evidence of ongoing systemic bacterial, fungal, or viral infection at the time of study enrollment visit
* Ongoing drug-induced liver injury, chronic active hepatitis B (HBV), alcoholic liver disease, non-alcoholic steatohepatitis, primary biliary cirrhosis, extrahepatic obstruction caused by cholelithiasis, cirrhosis of the liver, or portal hypertension.
* Ongoing alcohol or drug addiction
* Treatment with any other investigational agent or participating in another trial within 30 days prior to entering this study
* Breastfeeding or pregnancy
* Prior or ongoing clinically significant illness, medical condition, surgical history, physical finding, electrocardiogram (ECG) finding, or laboratory abnormality that, in the investigator's opinion, could adversely affect the safety of the subject or impair the assessment of study results.
* History of anaphylaxis in association with previous administration of monoclonal antibodies.
* Vaccination with a live vaccine within 28 days prior to start of therapy

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrolment:

* ECOG performance status >2
* History of a non-lymphoid malignancy except for the following: adequately treated local basal cell or squamous cell carcinoma of the skin, cervical carcinoma in situ, superficial bladder cancer, asymptomatic prostate cancer without known metastatic disease and with no requirement for therapy or requiring only hormonal therapy and with normal prostate specific antigen for ≥1 year prior to study enrollment visit, other Stage 1 or 2 cancer treated with a curative intent and currently in complete remission, for ≥3 years.
* Central nervous system lymphoma, leptomeningeal lymphoma, or histologic evidence of transformation to a high-grade or diffuse large B-cell lymphoma.
* Ann Arbor Stage I disease
* Ongoing immunosuppressive therapy other than corticosteroids
* Evidence of ongoing systemic bacterial, fungal, or viral infection at the time of study enrollment visit
* Ongoing drug-induced liver injury, chronic active hepatitis B (HBV), alcoholic liver disease, non-alcoholic steatohepatitis, primary biliary cirrhosis, extrahepatic obstruction caused by cholelithiasis, cirrhosis of the liver, or portal hypertension.
* Ongoing alcohol or drug addiction
* Treatment with any other investigational agent or participating in another trial within 30 days prior to entering this study
* Breastfeeding or pregnancy
* Prior or ongoing clinically significant illness, medical condition, surgical history, physical finding, electrocardiogram (ECG) finding, or laboratory abnormality that, in the investigator's opinion, could adversely affect the safety of the subject or impair the assessment of study results.
* History of anaphylaxis in association with previous administration of monoclonal antibodies.
* Vaccination with a live vaccine within 28 days prior to start of therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2018-11-23 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Complete Remission/Response (CR) rate | 24 weeks
  The complete Response rate (CR) is evaluated after the end of induction

SECONDARY OUTCOMES:
Progression free survival | 24 weeks
  Progression free survival (PFS) is defined as the time from registration to the first occurrence of progression or relapse as assessed by the investigator, or death from any cause. PFS for patients without disease progression, relapse, or death will be censored at the time of the last tumor assessment.
Overall survival | participants will be followed for their participation in the trial, an expected average of 8.6 years
  Overall survival is defined as the period from the induction registration to death from any cause. Patients who have not died until the time of the analysis will be censored at their last contact date.
Time to first response | participation will be followed for their participation in the trial, an expected average of 8.6 years
  Time to first response is defined as the time from the start of induction to first response (CR, PR).
Time to best response under treatment (induction and maintenance)Time | participation will be followed for their participation in the trial, an expected average of 8.6 years
  Time to best response is defined as the time from the start of induction to best response the patient achieves (CR, PR).
Response rate | 24 weeks
  The response rates (CR, PR) and overall response rate (CR, PR) are evaluated 4 weeks after the end of induction treatment.
Best response | participation will be followed for their participation in the trial, an expected average of 8.6 years
  Best response is determined in the time interval from the start of induction therapy to end of follow-up.
Time to Treatment failure | participation will be followed for their participation in the trial, an expected average of 8.6 years
  Time to treatment failure (TTF) is defined as the time of registration to discontinuation of therapy for any reason including death from any cause, progression, toxicity or add-on of new anti-cancer therapy. Patients alive without treatment failure are censored at the latest tumor assessment date.
Remission duration | participation will be followed for their participation in the trial, an expected average of 8.6 years
  Remission duration will be calculated in patients with response (CR, PR) to induction from end of induction to the date of progression, relapse or death from any cause. Patients alive without progression and relapse will be censored at the latest tumor assessment date or the stopping date.
Cause specific survival | participation will be followed for their participation in the trial, an expected average of 8.6 years
  Cause specific survival is defined as the period from the induction registration to death from lymphoma or lymphoma related cause; death unrelated to MZoL is considered as a competing event.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Buske, MD, Principal Investigator — University Hospital of Ulm
Locations (12):
- Germany (12):
  - Augusta-Kranken-Anstalt gGmbH, Bochum
  - University Hospital Essen, Essen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsmedizin Georg-August-University, Göttingen
  - University Hospital Halle, Halle
  - Institut für Versorgungsforschung GbR, Koblenz
  - University Hospital Mainz, Mainz
  - Universitätsklinikum Mannheim, Mannheim
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Münster
  - University Hospital Münster, Münster
  - Klinikum Passau, Passau
  - University Hospital Ulm, Ulm

REFERENCES:
- [Derived] Grunenberg A, Kaiser LM, Woelfle S, Schmelzle B, Viardot A, Moller P, Barth TF, Muche R, Dreyhaupt J, Buske C. Phase II trial evaluating the efficacy and safety of the anti-CD20 monoclonal antibody obinutuzumab in patients with marginal zone lymphoma. Future Oncol. 2020 May;16(13):817-825. doi: 10.2217/fon-2020-0071. Epub 2020 Mar 30. PMID 32223334